CLINICAL TRIAL: NCT04604821
Title: Delivering Enhanced Milieu Teaching (EM-Teach) Via Telehealth to Children and Families in Rural Communities
Brief Title: Delivering EMT Via Telehealth to Children and Families
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI decided to pursue the same aims using a different methodology, specifically a single-case experimental design, also called N-of-1 Trial to answer research questions after consultation with research mentors and consultants.
Sponsor: Oregon Health and Science University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Emily Quinn, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00019997
Record Dates: First submitted 2020-10-20; First posted 2020-10-27 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-02

CONDITIONS: Language Impairment
Keywords: Language Impairment; Telehealth; Rural; Enhanced Milieu Teaching
MeSH Terms: conditions — Language Disorders

STUDY DESIGN:
Intervention Model Description: Feasibility Study (Small Randomized Control Trial)
Who Masked: Outcomes Assessor
Masking Description: The assessor of the primary outcome will be blind to treatment condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Milieu Teaching (Experimental): Child-caregiver dyads receive up to 24 speech-language therapy sessions (50minutes, 2x per week for 3 months) where parents are taught by the interventionist to use Enhanced Milieu Teaching Strategies. Children and their families may continue to participate community-based educational programs.
  Interventions: Behavioral: Enhanced Milieu Teaching
- Community Treatment as Usual (Other): Child-caregiver dyads may continue to participate in community-based educational programs. Researchers provide up to 4 educational sessions to caregivers (50 minutes, every 3 weeks). During educational sessions parents are taught developmental milestones from the CDC Learn the Signs Act Early Public Health Campaign.
  Interventions: Behavioral: Parent Education

INTERVENTIONS:
Behavioral: Enhanced Milieu Teaching — A behavioral language intervention that uses naturally occurring interactions to facilitate young children's language skills.
  Arms: Enhanced Milieu Teaching
Behavioral: Parent Education — Parents receive information on child developmental milestones.
  Arms: Community Treatment as Usual

SUMMARY:
In the U.S., approximately 12% of children under 36 months have language impairments, yet less than 2% receive early language intervention. Early language intervention is underutilized nationally, with pronounced service gaps in rural communities. This gap is a significant issue because children with language impairments are at increased risk for learning and reading disabilities that can persist into adulthood. Telehealth has the potential to mitigate service gaps by improving access to treatments, increasing the availability of clinicians with expertise in language intervention, and reducing healthcare costs. Telehealth can alleviate logistic and geographic barriers to treatment facing children with disabilities and their families in rural communities. However, there is insufficient evidence on the effects of telehealth interventions for children with language impairments under 36 months. Consequently, there is an urgent need to explore innovative telehealth interventions with potential to improve the quality and efficiency of language treatments. The investigators will conduct a feasibility trial (small randomized control trial) to evaluate a telehealth intervention for children with language impairments and their caregivers.

DETAILED DESCRIPTION:
Aim 1: Explore stakeholders' preferences, experiences, and information needs regarding the delivery of language interventions via telehealth. Ethnographic interviews will be conducted with 16 stakeholders (n= 8 caregivers, 8 clinicians) to explore their preferences, experiences, and needs.

Aim 2: Determine the effect of telehealth Enhanced Milieu Teaching on caregiver language strategy use. Caregiver language strategy use will be compared between the intervention and control groups (n = 28 families, 14 intervention,14 control) during semi-structured caregiver-child interactions.

ELIGIBILITY:
Inclusion Criteria:

* (a) Child age between 18 and 36 months
* (b) developmental age of 9 months as measured on the Visual Reception Scale of the Mullen Scales of Early Learning (MSEL; 1995)
* (c) language delay as measured by a score of at least 1.33 SD below the mean on the Preschool Language Sclaes-5th Edition (PLS-5; Zimmerman, Steiner, & Evatt-Pond, 2011), and
* (d) hearing (with or without amplification) reported at 25dB HL or better confirmed by audiological testing, or medical record.

Exclusion Criteria:

* (a) primary diagnosis of any specific disability other than a language impairment including severe motor impairment
* (b) concomitant sensory impairments (e.g., hearing impairment, blindness), and
* (c) symptoms of autism spectrum disorder as measured by a result indicating "high risk" for autism (e.g., scores of 8 or higher) on the Modified Checklist for Autism In Toddlers-Revised with Follow-up (MCHAT-R/F Robins, Fein & Barton, 2009).

Ages: 18 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Parent use of EMT Strategies during a parent child interaction. | 1 pre-intervention assessment (start of study) and 1 post intervention assessment through study completion (3-4 months later).
  A parent-child interaction is a brief, repeatable, play-based, observational measure of a child's communicative performance during a 10-minute play period with the parent who agreed to participate in as a research volunteer in the study. It measures the number and percentage of correct of matched turns, expansions, time delays, and milieu teaching episodes during this play period.
  An increase in the Parent use of EMT strategies is a positive outcome.
  Metric/ Measurement Unit: Number and percentage of turns parents used EMT Strategies (e.g. matched turns, expansions, time delays, and milieu teaching episodes) during a 10 minute play interaction.

SECONDARY OUTCOMES:
Change in Productive Vocabulary on the Mac-Arthur Bates Communication Development Inventory (MCDI) score after 3-4 months of intervention | 1 pre-intervention assessment (start of study) and 1 post intervention assessment through study completion (3-4 months later).
  The MacArthur-Bates Communicative Development Inventory (MCDI) is a parent report instrument which captures important information about children's developing abilities in early language, including vocabulary comprehension, production, gestures, and grammar.
  An increase in the productive vocabulary represents a positive outcome.
  Metric/ Measurement Unit: Number of words expressed on the MCDI. The range of this instrument is 0 - 396.
Change in Individual Growth and Development Indicators for Infants and Toddlers- Early Communication Indicator (IGDI-ECI) score through 3-4 months of intervention | Once per month of intervention through study completion (3-4 months of intervention)
  The ECI is a brief, repeatable, play-based, observational measure of a child's communicative performance during a 6-minute play period with a familiar adult. It measures the number of gestures, vocalizations, single words, and multiple word combinations during this play period.
  An increase in the ECI presents a positive outcome.
  Metric/ Measurement Unit: Frequency count of communication utterances expressed during the 6 minute play interaction. ECI scores are weighted such that each single-word utterance is given a weight of two (each tally is multiplied by two), and each multiple word utterance is given a weight of three (each tally is multiplied by three)
Change in Preschool-Language Scales - 5th edition (PLS-5) | 1 pre-intervention assessment (start of study) and 1 post intervention assessment through study completion (3-4 months later).
  PLS™-5 Preschool Language Scales Fifth Edition offers a comprehensive developmental language assessment with items that range from pre-verbal, interaction-based skills to emerging language to early literacy.
  Increases on the PLS-5 represent a positive outcome.
  Metric/ Measurement Unit: Total Standard Score Range = 50 - 150 (Mean = 100, SD = 15).
  If we are unable to administer assessments to all participants in person due to public health impacts of COVID-19, we will report the raw scores because the PLS-5 is not standardized for telepractice administration. Raw scores range 0 - 132.
Change in number of Different Words on Structured Language Sample | 1 pre-intervention assessment (start of study) and 1 post intervention assessment through study completion (3-4 months later).
  A language sample is a naturalistic adult-child interaction with a specific set of toys to evaluate a child's spontaneous expressive language ability.
  Metric/ Measurement Unit: Change in frequency count of the number of different words spoken during a 20 minute language sample.

CONTACTS AND LOCATIONS:
Overall Officials: Emily D Quinn, Ph.D, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No